CLINICAL TRIAL: NCT02658565
Title: Surgical Staging for the Treatment of Endometrial Cancer Based on IOC
Brief Title: Selective Surgical Staging for the Treatment of Endometrial Cancer Based on Intraoperative Consultation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Frederick R. Ueland, M.D. (Other)
Responsible Party: Sponsor-Investigator, Frederick R. Ueland, M.D., Professor, Obstetrics and Gynecology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15-GYN-150
Record Dates: First submitted 2015-12-08; First posted 2016-01-20 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
Keywords: Intraoperative Consultation
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-risk for nodal involvement (No Intervention): No lymphadenectomy recommended
- High-risk for nodal involvement (Experimental): Lymphadenectomy recommended, including: obturator, iliac (internal, external, common) and aortic lymph nodes
  Interventions: Procedure: Lymphadenectomy

INTERVENTIONS:
Procedure: Lymphadenectomy — Lymphadenectomy recommended, including: obturator, iliac (internal, external, common) and aortic lymph nodes
  Arms: High-risk for nodal involvement

SUMMARY:
Complete pelvic and para-aortic lymphadenectomy performed at the time of primary surgical staging for endometrial cancer increases operative time and surgical morbidity, but appears to be necessary in most high grade and deeply invasive cancers. To date, the Mayo Clinic approach has not been reproduced, and the investigators propose to validate their algorithm at the University of Kentucky utilizing intra-operative consultation (IOC). The preliminary data at the University of Kentucky for IOC and endometrial cancer outcomes suggest that the investigators are well-suited to perform this investigation. A surgical approach that is tailored to the patient's cancer biology is rational, supported by the recent literature, and medically compelling since the co-morbidities of many obese, low-risk EC patients put them at significantly increased perioperative risk for complete lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be surgical candidates for complete hysterectomy and bilateral salpingo-oophorectomy and pelvic and aortic lymphadenectomy.
* Patients must have a histologically confirmed diagnosis of endometrial cancer and no clinical evidence of extra-uterine disease on preoperative evaluation.
* Preoperative evaluation to rule-out extra-uterine disease may include CT scan, MRI, or ultrasound. Preoperative imaging is not mandatory for study enrollment.
* Patients may have received prior systemic chemotherapy. Such therapy must have been completed at least 5 years prior to study entry and the patient has no evidence of disease subsequent to such therapy. Patients must not have received neoadjuvant chemotherapy for the present disease.
* Patients must have GOG performance status 0, 1, or 2.
* Patients must have an estimated survival greater than or equal to 3 months
* Patients must have signed an approved informed consent and HIPAA authorization.

Exclusion Criteria:

* Patients with clinical evidence of disease beyond the uterus, including presence of suspicious aortic or inguinal nodes on imaging or clinical exam.
* Patients who have received previous vaginal, pelvic, or abdominal irradiation.
* Patients who received chemotherapy directed at the present disease.
* Patients who have circumstances that will not permit completion of this study or the required follow-up.
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of surgical lymph node assessments.
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer within the last five years.
* Patients with GOG Performance Grade of 3 or 4.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 24 months
  Recurrence-free survival rates in low-risk and high-risk subgroups of patients with endometrial cancer as classified by the use of pathology intraoperative consultation (IOC).

SECONDARY OUTCOMES:
Progression-free survival | 5 years
  Progression-free survival rates in low-risk and high-risk subgroups of patients with endometrial cancer as classified by the use of pathology intraoperative consultation (IOC)
Disease-specific Survival | 5 years
  Disease-specific survival rates in low-risk and high-risk subgroups of patients with endometrial cancer as classified by the use of pathology intraoperative consultation (IOC)
Overall patient survival | 5 years
  Overall survival rates in low-risk and high-risk subgroups of patients with endometrial cancer as classified by the use of pathology intraoperative consultation (IOC)
Concordance between IOC and final pathology Incidence | 5 years
Perioperative morbidity and mortality | 5 years
  Perioperative morbidity and mortality outcome will be assessed as the number of participants with Adverse Events/death which are related to treatment/surgery .

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Ueland, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No